CLINICAL TRIAL: NCT03742206
Title: Comparison of Parasacral Transcutaneous Electrical Stimulation With Transcutaneous Posterior Tibial Nerve Stimulation in Women With Overactive Bladder: a Randomized Clinical Trial
Brief Title: Comparison of Two Forms of Transcutaneous Electrical Stimulation in Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-0056
Record Dates: First submitted 2018-10-31; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Overactive Bladder; Urinary Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parasacral (Experimental): Parasacral Transcutaneous Electrical Stimulation Group: participants in this group will receive two self-adhesive electrodes and will be instructed to position them in the sacral region. Current parameters will be: 10 hertz frequency, 700μs wavelength, 20 minute therapy duration, 3x frequency in the week. The treatment will be at home for 6 weeks.
  Interventions: Device: Parasacral Transcutaneous Electrical Stimulation
- Posterior Tibial Nerve (Active Comparator): Transcutaneous Posterior Tibial Nerve Stimulation Group: participants in this group will receive a neoprene ankle brace that will be connected to the electrostimulator. Current parameters will be: 10 hertz frequency, 700μs wavelength, 20 minute therapy duration, 3x frequency in the week. The treatment will be at home for 6 weeks.
  Interventions: Device: Transcutaneous Posterior Tibial Nerve Stimulation

INTERVENTIONS:
Device: Parasacral Transcutaneous Electrical Stimulation — Electrical stimulation with surface electrodes on the sacral roots of S3 that produce inferior urinary tract neuromodulation.
  Arms: Parasacral
Device: Transcutaneous Posterior Tibial Nerve Stimulation — Electrical stimulation with surface electrodes through the activation of peripheral afferent nerves that produce inferior urinary tract neuromodulation
  Arms: Posterior Tibial Nerve

SUMMARY:
Aim: To compare the effects of parasacral transcutaneous electrical stimulation with transcutaneous posterior tibial nerve stimulation on the symptoms of Overactive Bladder in women.

Study's hypothesis: The use of the parasacral transcutaneous electrical stimulation technique presents better results regarding the remission of overactive bladder symptoms in relation to transcutaneous posterior tibial nerve stimulation.

DETAILED DESCRIPTION:
Search location: The data will collected at the Ambulatory of Urogynecology and Obstetrics of Porto Alegre Clinical Hospital (HCPA), where the activities of Pelvic Physiotherapy are performed

Main outcome: to measure changes in urinary urgency and quality of life.

Secondary outcome: to measure changes in the severity of urinary incontinence and the symptom bother.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of overactive bladder with or without the presence of urinary incontinence.
* Understand the instruments used in the research.

Exclusion Criteria:

* Urinary tract infection
* Neurological disease
* Other previous treatment in the last four weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment in quality of life | six weeks
  Application of the King's Health Questionnaire (KHQ). KHQ is an instrument for measuring quality of life in people diagnosed with urinary incontinence, consisting of 30 objective questions distributed in 9 domains. In each question, values are assigned according to the intensity of the patient's complaint (0 = not applicable, 1 = no; 2 = a little / sometimes, 3 = more or less / several times, 4 = a lot / always). The final score is calculated individually for each domain and ranges from 0 to 100, the highest score being related to a poorer quality of life.

SECONDARY OUTCOMES:
Severity of urinary incontinence | six weeks
  Application of the Incontinence Severity Index. It is a brief instrument, consisting of two questions regarding the frequency and amount of urinary loss. The final score obtained by multiplying the frequency scores by the amount of urinary loss allows the incontinence urinary to be classified as mild (final score 1-2), moderate (final score 3-6 ), severe (final score 8-9) and very severe (final score 12).
Severity of overactive bladder symptoms | six weeks
  Application of the Symptom Bother Scale. It instrument asks how bothered the patient is by the 4 hallmark symptoms of overactive bladder: urinary frequency, urgency, nocturia, and urge incontinence. Patients respond on a 6-point Likert scale ranging from 0 (not at all) to 5 (a very great deal), with a maximum possible score of 40, calculated by adding all responses.

CONTACTS AND LOCATIONS:
Overall Officials: José Geraldo Lopes Ramos, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Suzana Mallmann, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided